CLINICAL TRIAL: NCT06963489
Title: Cerebral Large Vessel Occlusion Stroke Multiomics Biosample Cohort
Acronym: CLOMB
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Beijing Tiantan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Baotou Central Hospital (Other); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jie Xu, Deputy Director, First Affiliated Hospital of Wannan Medical College
Other Study IDs: 202543
Record Dates: First submitted 2025-04-28; First posted 2025-05-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Large Vessel Occlusion; Acute Ischemic Stroke
Keywords: multiomics; acute ischemic stroke with large vessel occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — intracranial thrombi, intracranial occluded segment blood, peripheral arterial blood, peripheral venous blood,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — Intervention is not applicable

SUMMARY:
This multicenter, ambispective cohort study establishes a comprehensive multiomics biobank from five stroke centers, encompassing thrombi, intracranial blood, peripheral arterial/venous blood, and clinical-laboratory-imaging-follow-up data from patients with acute ischemic stroke with large vessel occlusion (AIS-LVO).

DETAILED DESCRIPTION:
This study is a multicenter, ambispective cohort study. Blood clot, peripheral arterial blood, peripheral venous blood, and intracranial blood samples were collected from patients at 5 stroke centers to establish a biobank of patients with AIS-LVO.

Blood and thrombus samples underwent pathological analysis, metabolomics, proteomics, and genomics for multidimensional testing. Additionally, clinical, laboratory, follow-up, and imaging data were collected.

The main objective is to identify phenotypic differences between intracranial blood and peripheral blood, describe the microenvironment profile, and perform a combined analysis of the thrombus' multi-omics phenotypes to construct a "microenvironment" multiomics fingerprint.

Furthermore, based on the multi-omics phenotypic components of thrombus and blood, clinical prediction models will be built. These models will address clinical issues related to etiology diagnosis, risk stratification, and prognosis in large vessel occlusion stroke patients, using external or internal validation methods.

For a subset of patients, thrombus samples will undergo pathological processing and histological examination, followed by joint analysis with multi-omics data.

The CLOMB study was designed to collect multidimensional clinical and multiomics data of AIS-LVO patients. The rich data set with deep phenotypes and multiomics analysis of patients will facilitate the study of more stroke-related scientific questions, which include but not limit to the following:

1. Thrombus and microenvironment multiomics profiles
2. Identification of post-stroke therapeutic target
3. Establishing new prediction and risk stratification models based on multiomics data
4. Exploring new diagnostic approach for AIS-LVO etiologies

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Patients with intracranial and extracranial large vessel occlusion ischemic stroke confirmed by cerebrovascular angiography.
3. Availability of complete clinical and follow-up information required for the study.
4. Availability of blood and/or thrombus biological samples.
5. Voluntary written informed consent signed by the patient or their family (1) For retrospectively enrolled patients, a "broad informed consent" was signed at the time of sample collection. Upon enrollment into the cohort, a follow-up phone call was made to confirm the informed consent.

(2) For prospectively enrolled patients, informed consent for this study was signed at the time of enrollment by the patient or their family.

Exclusion Criteria:

1. Patients for whom biological samples cannot be obtained;
2. Patients or their family members who refuse to sign the informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We include patients with acute large vessel occlusion ischemic stroke from at least 5 stroke centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Number of patients with futile recanalization | From enrollment to 3 month follow-up
  mRS score ≥3 at 3 months

SECONDARY OUTCOMES:
Number of patients with specific stroke etiologies | Baseline
  Patients will be classified as Cardioembolism or Large artery atherosclerosis as a final stroke etiology.
Number of patients with hemorrhagic transformation | 7 days within stroke onset
  HT: secondary occurrence of bleeding within an area of the brain affected by ischemic stroke (cerebral infarction).
  Further stratified into:
  1. symptomatic intracranial hemorrhage (sICH) and asymptomatic intracranial hemorrhage (aICH)
  2. different extent: HI1, HI2, PH1, PH2
Number of patients with infarct expansion | Baseline
  Patients undergoing thrombectomy had their CTAVP reexamined 24 hours later. Through CTP, it was determined whether the volume of the infarcted lesion (rCBF<30%) had expanded compared with preoperative CTP.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The First Affiliated Hospital of Shihezi University, Wuhu, Anhui
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine Hospital, Jinan, Shandong
  - The First Affiliated Hospital of zhengzhou University, Henan, Zhengzhou
  - Capital medical university of Beijing Tiantan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu X, Song Y, Cao W, Bai X, Wang X, Gao P, Chen J, Chen Y, Yang B, Wang Y, Chen F, Ma Q, Yu B, Jiao L. Alterations of Hemostatic Molecular Markers During Acute Large Vessel Occlusion Stroke. J Am Heart Assoc. 2024 Feb 6;13(3):e032651. doi: 10.1161/JAHA.123.032651. Epub 2024 Jan 31. PMID 38293908
- [Background] Kollikowski AM, Schuhmann MK, Nieswandt B, Mullges W, Stoll G, Pham M. Local Leukocyte Invasion during Hyperacute Human Ischemic Stroke. Ann Neurol. 2020 Mar;87(3):466-479. doi: 10.1002/ana.25665. Epub 2020 Jan 16. PMID 31899551
- [Background] Strinitz M, Pham M, Marz AG, Feick J, Weidner F, Vogt ML, Essig F, Neugebauer H, Stoll G, Schuhmann MK, Kollikowski AM. Immune Cells Invade the Collateral Circulation during Human Stroke: Prospective Replication and Extension. Int J Mol Sci. 2021 Aug 25;22(17):9161. doi: 10.3390/ijms22179161. PMID 34502070
- [Background] Stoll G, Schuhmann MK, Nieswandt B, Kollikowski AM, Pham M. An intravascular perspective on hyper-acute neutrophil, T-cell and platelet responses: Similarities between human and experimental stroke. J Cereb Blood Flow Metab. 2022 Sep;42(9):1561-1567. doi: 10.1177/0271678X221105764. Epub 2022 Jun 8. PMID 35676801
- [Background] Zimmermann L, Pham M, Marz AG, Kollikowski AM, Stoll G, Schuhmann MK. Defining cerebral leukocyte populations in local ischemic blood samples from patients with hyperacute stroke. J Cereb Blood Flow Metab. 2022 May;42(5):901-904. doi: 10.1177/0271678X221078617. Epub 2022 Feb 2. PMID 35107055
- [Background] Dargazanli C, Blaquiere M, Moynier M, de Bock F, Labreuche J, Ter Schiphorst A, Derraz I, Radu RA, Gascou G, Lefevre PH, Rapido F, Fendeleur J, Arquizan C, Bourcier R, Marin P, Machi P, Cagnazzo F, Hirtz C, Costalat V, Marchi N. Inflammation biomarkers in the intracranial blood are associated with outcome in patients with ischemic stroke. J Neurointerv Surg. 2025 Jan 17;17(2):159-166. doi: 10.1136/jnis-2023-021365. PMID 38514190
- [Background] Costamagna G, Bonato S, Corti S, Meneri M. Advancing Stroke Research on Cerebral Thrombi with Omic Technologies. Int J Mol Sci. 2023 Feb 8;24(4):3419. doi: 10.3390/ijms24043419. PMID 36834829
- [Background] Staessens S, Fitzgerald S, Andersson T, Clarencon F, Denorme F, Gounis MJ, Hacke W, Liebeskind DS, Szikora I, van Es A, Brinjikji W, Doyle KM, De Meyer SF. Histological stroke clot analysis after thrombectomy: Technical aspects and recommendations. Int J Stroke. 2020 Jul;15(5):467-476. doi: 10.1177/1747493019884527. Epub 2019 Nov 3. PMID 31679478
- [Background] Staessens S, Francois O, Brinjikji W, Doyle KM, Vanacker P, Andersson T, De Meyer SF. Studying Stroke Thrombus Composition After Thrombectomy: What Can We Learn? Stroke. 2021 Nov;52(11):3718-3727. doi: 10.1161/STROKEAHA.121.034289. Epub 2021 Sep 14. PMID 34517770
- [Background] Patil S, Darcourt J, Messina P, Bozsak F, Cognard C, Doyle K. Characterising acute ischaemic stroke thrombi: insights from histology, imaging and emerging impedance-based technologies. Stroke Vasc Neurol. 2022 Aug;7(4):353-363. doi: 10.1136/svn-2021-001038. Epub 2022 Mar 3. PMID 35241632
- [Background] Widimsky P, Snyder K, Sulzenko J, Hopkins LN, Stetkarova I. Acute ischaemic stroke: recent advances in reperfusion treatment. Eur Heart J. 2023 Apr 7;44(14):1205-1215. doi: 10.1093/eurheartj/ehac684. PMID 36477996